CLINICAL TRIAL: NCT02167763
Title: Study of the VeraCept Intrauterine Device for Long Acting Reversible Contraception
Brief Title: Comparative Study of the VeraCept Low-Dose Intrauterine Copper Contraceptive vs. the TCu380 Copper IUD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CM2010.01
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Prevention of Pregnancy
Keywords: contraception; IUD; copper

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- VeraCept Intrauterine Contraceptive (Experimental): The VeraCept low-dose Intrauterine Copper Contraceptive
  Interventions: Device: VeraCept Intrauterine Copper Contraceptive
- TCu380 (Active Comparator): A commercial standard T-shaped copper IUD (TCu380)
  Interventions: Device: TCu380 IUD

INTERVENTIONS:
Device: VeraCept Intrauterine Copper Contraceptive
  Arms: VeraCept Intrauterine Contraceptive
Device: TCu380 IUD
  Arms: TCu380

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the VeraCept Low Dose Intrauterine Copper Contraceptive compared to the standard T shaped copper IUD, the TCu380.

DETAILED DESCRIPTION:
This is a prospective, randomized, subject-blinded, two arm controlled study of the Safety, Feasibility and Effectiveness of the VeraCept low-dose intrauterine copper contraceptive as compared to a concurrently controlled, commercially available standard copper "T" IUD (TCu380).

ELIGIBILITY:
Inclusion Criteria:

* Adult females ages 18 to 42 (pre-menopausal)
* Have had at least one child (parous) and currently seeking long acting reversible contraception
* Normal uterine cavity as determined by ultrasound
* Willing to sign informed consent
* Able and willing to comply with study assessment schedule

Exclusion Criteria:

* Post menopausal
* Pregnant (at time of enrollment)
* Known anatomical abnormalities of uterus, cervix and/or fallopian tubes
* Diagnosed or in treatment for cancer
* Untreated acute cervicitis
* In treatment for active Pelvic Inflammatory Disease
* Unexplained uterine bleeding or menometrorrhagia
* Known allergy to copper (Wilson's Disease) or imaging contrast media
* Unsuitable for study participation in the opinion of the Principal Investigator

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Contraceptive Effectiveness | 12 Months
  Number of subjects who become pregnant during the study period
Placement Feasibility | At Enrollment
  Ability of the clinician to successfully place the device

SECONDARY OUTCOMES:
Device Expulsion | 12 Months
  Number of subjects identified with partially or fully expelled devices
Tolerability | 12 Months
  Number of subjects who request device removal due to inability to tolerate the intervention (device)
Pain at Insertion | At Enrollment
  Subject reported pain scores at device insertion

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. Canela, M.D., Principal Investigator — Clinica Canela
Locations (1):
- Clinica Canela, La Romana, Dominican Republic